CLINICAL TRIAL: NCT00611923
Title: Androgen Hormones in PMDD
Brief Title: Effectiveness of Flutamide in Treating Women With Premenstrual Dysphoric Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R34MH072878 (NIH); R34MH072878 (NIH); DATR A5-ETPD
Record Dates: First submitted 2008-02-06; First posted 2008-02-11 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Dysphoric Disorder; PMDD; PMS
MeSH Terms: conditions — Premenstrual Syndrome; Premenstrual Dysphoric Disorder | interventions — Flutamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- B (Placebo Comparator): Participants will take placebo flutamide
  Interventions: Drug: Placebo
- A (Experimental): Participants will take flutamide
  Interventions: Drug: Flutamide

INTERVENTIONS:
Drug: Flutamide — Participants will take one 125-mg flutamide capsule twice a day for two menstrual cycles. If a participant is unable to tolerate a twice-daily dose due to side effects, the dose will be reduced to one capsule per day.
  Other Names: Eulexin
  Arms: A
Drug: Placebo — Participants will take a lactose capsule twice a day for two menstrual cycles. If a participant is unable to tolerate a twice-daily dose due to side effects, the dose will be reduced to one capsule per day.
  Arms: B

SUMMARY:
This study will evaluate the effectiveness of flutamide in reducing symptoms of premenstrual dysphoric disorder.

DETAILED DESCRIPTION:
Premenstrual dysphoric disorder (PMDD) is a condition that affects about 5% of menstruating women. Women with PMDD experience serious emotional and physical disturbances, which may include depression, tension, irritability, anger, anxiety, and sleep and appetite problems. Symptoms of PMDD are directly linked with the menstrual cycle, generally beginning in the latter half of the cycle and ending around the start of the next cycle. If left unmanaged, PMDD may interfere with a woman's ability to carry out normal day-to-day functioning. Current treatments for PMDD include medications, psychotherapy, and nutritional modifications. Flutamide, a medication that blocks the action of testosterone and other mood-influencing hormones, may be helpful in alleviating symptoms of PMDD. This study will evaluate the effectiveness of flutamide in reducing symptoms of premenstrual dysphoric disorder.

This two-phase study will last a total of 4 months and will include 7 study visits. Phase 1 will last 2 months and will include Visits 1 through 3. During Phase 1, participants will keep a daily record of symptoms, participate in a diagnostic interview, and undergo a medical history review, a physical exam, and screening laboratory tests. Eligible participants will then enter Phase 2, the treatment phase of the study.

During the treatment phase, participants will be randomly assigned to take flutamide or placebo for 2 months. Study visits will occur every 2 weeks and will include Visits 4 through 7. These visits will include discussion of side effects, symptom rating, and laboratory tests to check for pregnancy and any side effects related to liver function, blood counts, or blood chemistry. At the end of treatment with flutamide or placebo, participants will have the option of receiving treatment with sertraline, an antidepressant known to be effective for many women with PMDD. Sertraline will be given during the 2 premenstrual weeks for two cycles. If participants have already unsuccessfully tried sertraline for PMDD treatment, an alternative treatment can be attempted.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for PMDD by history
* Regular menstrual cycles that are 25 to 35 days in length during the year prior to study entry
* Willing to use barrier methods of birth control during the study if sexually active
* If engaged in psychotherapy for at least 3 months before study entry, participation will be allowed if the intensity of psychotherapy remains the same during the study
* Normal PAP and physical exam, including pelvic exam, within the 1 year prior to study entry

Exclusion Criteria:

* Use of oral contraceptives or other exogenous hormone preparations within the 3 months prior to study entry
* Suicide attempt or severe suicidal ideation within the 2 years prior to study entry
* History of any psychotic disorder or bipolar disorder
* Substance abuse, except nicotine, within the 6 months prior to study entry
* Use of pharmacological treatment for PMDD symptoms (e.g., antidepressants, hormones, gonadotropin-releasing hormone agonists, anxiolytics, calcium, herbal preparations, diuretics) within the 3 months prior to study entry
* Daily use of psychotropic or anticonvulsant medications within the 3 months prior to study entry
* Use of sleeping pills more than once per week
* Consumption of more than 50 ounces of alcohol per week
* Pregnant or breastfeeding
* Hepatic, renal, autoimmune, or chronic inflammatory disease
* Seizure disorder
* Inability to read or follow instructions in English

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2005-02; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Altemus, MD, Principal Investigator — Weill Medical College of Cornell University

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 115 subjects enrolled in the screening phase of the study. 27 subjects qualified for randomization and 25 of those agreed to participate in the treatment study.
Groups:
- Placebo: Participants will take placebo flutamide
  Placebo: Participants will take a lactose capsule twice a day for two menstrual cycles. If a participant is unable to tolerate a twice-daily dose due to side effects, the dose will be reduced to one capsule per day.
- Flutamide: Participants will take flutamide
  Flutamide: Participants will take one 125-mg flutamide capsule twice a day for two menstrual cycles. If a participant is unable to tolerate a twice-daily dose due to side effects, the dose will be reduced to one capsule per day.
Period: Overall Study
Arm/Group | Placebo | Flutamide
Started | 12 | 13
Completed | 10 | 11
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Flutamide | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Full Range); unit: years] | 34.3 [21 to 50] | 36.3 [23 to 44] | 35.3 [21 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 12 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Premenstrual Symptoms as Measured by the Premenstrual Tension Scale (PMTS)
Description: Low score on PMTS scale is 0 and high score is 40. Change score is calculated as PMTS score at month 1 or month 2 minus baseline PMTS score. Negative change score is a reduction in symptoms during treatment and positive change score is an increase in symptoms during treatment.
Time Frame: Measured at Months 1and 2
Population: 12 subjects were randomized to placebo and 13 randomized to flutamide. At the one month visit 11 subjects taking placebo and 13 subjects taking flutamide provided PMTS ratings. At the two month visit 10 subjects taking placebo and 11subjects randomized to flutamide provided PMTS ratings
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Flutamide
Number analyzed (Participants) | 11 | 13
score on a scale
  Month 1 | -6.9 (2.3) | -5.5 (2.1)
  Month 2: number analyzed (Participants) | 10 | 11
  Month 2 | -5.5 (2.2) | -8.3 (2.1)
Statistical Analysis 1: Comparison: Placebo vs Flutamide; paired t-test analysis comparing change from baseline PMTS score at month 1 between flutamide and placebo groups; Test type: Superiority or Other; p = 0.57, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Flutamide; paired t-test analysis comparing change from baseline PMTS score at month 2 between flutamide and placebo groups; Test type: Superiority or Other; p = .27, t-test, 2 sided

2. Secondary Outcome: Change in Premenstrual Symptoms as Measured by the Daily Rating of Severity of Problems (DRSP) Scale
Description: DRSP low score is 21 high score is 126. High score indicates more severe symptoms. Average score for the 4 days preceding menses was calculated for each subject in each cycle. Change score is calculated as DRSP score at month 1 or month 2 minus baseline DRSP score. Negative change score is a reduction in symptoms during treatment and positive change score is an increase in symptoms during treatment.
Time Frame: Measured at Months 1 and 2
Population: 12 subjects were randomized to placebo and 13 randomized to flutamide. At the one month visit 10 subjects taking placebo and 12 subjects taking flutamide provided DRSP ratings. At the two month visit 10 subjects taking placebo and 12 subjects randomized to flutamide provided DRSP ratings
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Flutamide
Number analyzed (Participants) | 10 | 12
score on a scale
  Month 1 | -21.3 (5.3) | -26.0 (4.9)
  Month 2 | -22.2 (7.5) | -35.6 (6.8)
Statistical Analysis 1: Comparison: Placebo vs Flutamide; paired t-test comparing change in DRSP scores from baseline to Month 1 of treatment Larger positive change score indicates a greater reduction in symptoms from baseline; Test type: Superiority or Other; p = 0.52, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Flutamide; paired t-test comparing change in DRSP scores from baseline to Month 2 of treatment Larger positive change score indicates a greater reduction in symptoms from baseline; Test type: Superiority or Other; p = 0.2, t-test, 2 sided

3. Secondary Outcome: Side Effect Burden Measured by Side Effect Questionnaire
Description: The Side Effects Questionnaire is a measure of combined side effect burden, including a score for frequency (0-6), intensity (0-6) and interference with function (0-6). Low score is 0, high score is 18, High score represents greater severe side effect burden
Time Frame: Measured at Months 1 and 2
Population: 12 subjects were randomized to placebo and 13 randomized to flutamide. At the one month visit 11 subjects taking placebo and 13 subjects taking flutamide provided side effect ratings. At the two month visit 10 subjects taking placebo and 10 subjects randomized to flutamide provided side effect ratings
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Flutamide
Number analyzed (Participants) | 11 | 13
score on a scale
  Month 1 | 3.9 (1.4) | 3.5 (1.3)
  Month 2: number analyzed (Participants) | 10 | 10
  Month 2 | 2.2 (1.2) | 5.1 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Flutamide; Test type: Superiority or Other; p = 0.8, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Flutamide; Test type: Superiority or Other; p = 0.1, t-test, 2 sided

4. Secondary Outcome: Premenstrual Symptoms as Measured by the Clinical Global Improvement Scale at Month 1 and Month 2
Description: Scale range in 1-7. 1 is very much improved compared to baseline, 4 is no change compared to baseline, and 7 is very much worse compared to baseline.
Time Frame: Measured at Months 1 and 2
Population: 12 subjects were randomized to placebo and 13 randomized to flutamide. At the one month visit 11 subjects taking placebo and 13 subjects taking flutamide had CGI-improvement ratings. At the two month visit 10 subjects taking placebo and 12 subjects randomized to flutamide had CGI-improvement ratings
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Flutamide
Number analyzed (Participants) | 11 | 13
score on a scale
  Month 1 | 3.2 (0.3) | 2.5 (0.3)
  Month 2: number analyzed (Participants) | 10 | 12
  Month 2 | 3.1 (0.3) | 2.2 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Flutamide; paired t-test was performed comparing the Clinical Global Improvement score at month 1 between placebo and flutamide groups; Test type: Superiority or Other; p = .15, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Flutamide; t-test was performed comparing the Clinical Global Improvement score at month 2 between placebo and flutamide groups; Test type: Superiority or Other; p = .05, t-test, 2 sided

5. Other Pre Specified Outcome: Change in Clinical Global Severity Scale
Description: Scale range in 1-7. 1 is not at all ill, 4 is moderately ill, and 6 is severely ill and 7 is among the most extremely ill patients. Change score is calculated as Clinical Global Severity Scale score at the end of treatment month 1 or treatment month 2 minus baseline score. Negative change score is a reduction in symptoms during treatment and a positive change score is an increase in symptoms during treatment.
Time Frame: Measured at Month 1 and Month 2
Population: 12 subjects were randomized to placebo and 13 randomized to flutamide. At the one month visit 11 subjects taking placebo and 13 subjects taking flutamide provided CGI severity ratings. At the two month visit 10 subjects taking placebo and 11subjects randomized to flutamide provided CGI severity ratings
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Flutamide
Number analyzed (Participants) | 11 | 13
score on a scale
  Month 1 | -0.9 (0.4) | -1.2 (0.4)
  Month 2: number analyzed (Participants) | 10 | 11
  Month 2 | -0.5 (0.4) | -1.7 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Flutamide; Test type: Superiority or Other — Comparison of change from baseline score to treatment month 1 between placebo and flutamide treated subjects; p = 0.5, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Flutamide; Test type: Superiority or Other — paired t-test analysis comparing change from baseline CGI severity score at month 2 between flutamide and placebo groups; p < .04, t-test, 2 sided

6. Other Pre Specified Outcome: Change in Premenstrual Symptoms as Measured by the Patient Global Premenstrual Symptoms as Measured by the Patient Global Improvement Scale at Month 1 and Month 2
Description: Scale range in 1-7. 1 is very much improved, 4 is no change, and 7 is very much worse.
Time Frame: Measured at Month 1 and Month 2
Population: 12 subjects were randomized to placebo and 13 randomized to flutamide. At the one month visit 11 subjects taking placebo and 12 subjects taking flutamide had Patient Global Improvement Scale ratings. At the two month visit 10 subjects taking placebo and 11 subjects randomized to flutamide had Patient Global Improvement Scale ratings
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Flutamide
Number analyzed (Participants) | 11 | 12
score on a scale
  Month 1 | 3.0 (0.3) | 2.4 (0.3)
  Month 2: number analyzed (Participants) | 10 | 11
  Month 2 | 2.2 (0.3) | 3.1 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Flutamide; paired t-test was performed comparing the Patient Global Improvement score at month 1 between placebo and flutamide groups; Test type: Superiority or Other; p = 0.2, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Flutamide; Test type: Superiority or Other — paired t-test was performed comparing the Patient Globall Improvement score at treatment month 2 between placebo and flutamide groups; p = 0.06, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 months per subject
Description: One subject randomized to placebo never took the medication after it was dispensed, so is not included in the adverse event table.
Arm/Group | Placebo | Flutamide
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 7/11 | 11/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | Flutamide (N=13)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
hot flushes (Vascular disorders) | 0 (0) | 2 (2)
headache (Nervous system disorders) | 1 (1) | 5 (5)
parasthesia (Nervous system disorders) | 0 (0) | 1 (1)
stomach pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
insomnia (Nervous system disorders) | 2 (2) | 2 (2)
leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
dry mouth (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
fatigue (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes